CLINICAL TRIAL: NCT03296228
Title: Comparison of Dynamic Radiographs in Determining Fusion Level in Adolescent Idiopathic Scoliosis Correction
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Collaborators: AO Foundation, AO Spine (Other)
Responsible Party: Principal Investigator, Dr. Kenny Kwan, Clinical Assistant Professor, The University of Hong Kong
Other Study IDs: UW 16-208
Record Dates: First submitted 2017-09-22; First posted 2017-09-28 (Actual); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Adolescent Idiopathic Scoliosis
Keywords: AIS
MeSH Terms: interventions — Supine Position

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hong Kong: Radiation: Flexibility Radiographs (supine, supine side-bend, FB)
  supine side-bending and fulcrum bending films
  Interventions: Radiation: Flexibility Radiographs (supine, supine side-bend, FB)
- Turkey: Radiation: Flexibility Radiographs (supine, supine side-bend, FB)
  Radiation: Flexibility Radiographs (awake traction)
  Radiation: Flexibility Radiographs (STUGA)
  supine side-bending, fulcrum bending films, awake traction and supine traction under GA
  Interventions: Radiation: Flexibility Radiographs (supine, supine side-bend, FB); Radiation: Flexibility Radiographs (awake traction); Radiation: Flexibility Radiographs (STUGA)

INTERVENTIONS:
Radiation: Flexibility Radiographs (supine, supine side-bend, FB) — Supine, supine side-bend, fulcrum bend
Radiation: Flexibility Radiographs (awake traction) — awake traction
  Groups: Turkey
Radiation: Flexibility Radiographs (STUGA) — supine traction under GA
  Groups: Turkey

SUMMARY:
The purpose of this study is to identify the flexibility radiograph(s) that can most accurately predict the curve behaviour after surgical correction of AIS. With these findings, the investigators hope to give further guidance for the selection of fusion levels and to incorporate different dynamic radiographs into the Lenke Classification, leading to a more universal application that can consistently lead to good surgical and clinical outcome.

DETAILED DESCRIPTION:
The Lenke Classification is the most widely-accepted classification for Adolescent Idiopathic Scoliosis (AIS) in the world. Its recommendations for fusion of the minor curves depend on its structurality. It defines a minor curve as structural if there is inflexibility on side-bending more than 25 . However, a recent Delphi survey from a panel of experts in AIS management showed that there was no consensus as to which type of dynamic radiograph was optimal. Up to two thirds of the surgeons did not use side-bending as a routine, and hence they cannot apply the Lenke Classification accurately in clinical practice nor follow its recommendations for fusion.

Furthermore, the current classification does not give specific recommendations regarding the selection of fusion levels and does not take into account the clinical appearance of the patients which impact on treatment. Consequently, there are still controversies regarding the Upper Instrumented Vertebra (UIV) and Lowest Instrumented Vertebra (LIV) selections, and following the recommendations may not allow fusion of the least number of segments nor give best clinical results eg shoulder balance.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with AIS who reach the threshold for surgical correction.
* Patients aged 10 to 18 years

Exclusion Criteria:

* Neuromuscular deformity
* Prior fusion or spine surgery
* Spinal tumor diagnosis
* Congenital anomalies

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study will be divided into two phases. In Phase 1, an exploratory pilot study will be performed with up to 3 flexibility films done on the same patient in different spinal centres which are in Hong Kong and Turkey.
Sampling Method: Non-Probability Sample
Enrollment: 134 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Investigate the flexibility equivalence of different bending methods, and their predictability of the final outcome | 6 months to 9 months
  To investigate the flexibility equivalence of different bending methods: supine side-bending, fulcrum bending (FB) and supine Halter traction without GA (awake), and their predictability of the final outcome

SECONDARY OUTCOMES:
Incorporate these findings into the Lenke Classification of AIS | 6 months to 9 months
  To incorporate these findings into the Lenke Classification of AIS
Give new recommendations for fusion levels according to the flexibility assessment | 6 months to 9 months
  To give new recommendations for fusion levels according to the flexibility assessment

CONTACTS AND LOCATIONS:
Overall Officials: Dr Kenny Kwan, BMBCh(Oxon), Principal Investigator — The University of Hong Kong
Locations (1):
- Duchess of Kent Children's Hospital, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hamzaoglu A, Talu U, Tezer M, Mirzanli C, Domanic U, Goksan SB. Assessment of curve flexibility in adolescent idiopathic scoliosis. Spine (Phila Pa 1976). 2005 Jul 15;30(14):1637-42. doi: 10.1097/01.brs.0000170580.92177.d2. PMID 16025034
- [Background] Clements DH, Marks M, Newton PO, Betz RR, Lenke L, Shufflebarger H; Harms Study Group. Did the Lenke classification change scoliosis treatment? Spine (Phila Pa 1976). 2011 Jun 15;36(14):1142-5. doi: 10.1097/BRS.0b013e318207e9c4. PMID 21358471
- [Background] Cheh G, Lenke LG, Lehman RA Jr, Kim YJ, Nunley R, Bridwell KH. The reliability of preoperative supine radiographs to predict the amount of curve flexibility in adolescent idiopathic scoliosis. Spine (Phila Pa 1976). 2007 Nov 15;32(24):2668-72. doi: 10.1097/BRS.0b013e31815a5269. PMID 18007242
- [Background] Lenke LG, Betz RR, Harms J, Bridwell KH, Clements DH, Lowe TG, Blanke K. Adolescent idiopathic scoliosis: a new classification to determine extent of spinal arthrodesis. J Bone Joint Surg Am. 2001 Aug;83(8):1169-81. PMID 11507125
- [Background] Chow SC, Shao J, Wang H. Sample Size Calculations in Clinical Research. 2003. Marcel Dekker, New York